CLINICAL TRIAL: NCT03101397
Title: The Clinical Value of Serum KL-6 Changes on Evaluating Disease Development in Different Diffuse Parenchymal Lung Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, chen miao, Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: gyfyy-2017
Record Dates: First submitted 2017-03-23; First posted 2017-04-05 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Diffuse Parenchymal Lung Disease
Keywords: serum KL-6; pulmonary function test; CT score; evaluation
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood biomakers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- improved group: defined by two or more of the following: A decrease in symptoms, specifically an increase in the level of exertion required before the patient must stop because of breathlessness or a decline in the frequency or severity of cough Reduction of parenchymal abnormalities on chest CT scan Physiologic improvement defined by > 10% increase in FVC (or at least > 200-ml change) or > 15% increase in single-breath DLCO (or at least > 3 ml/min/mm Hg)
- deteriorated group: defined by two or more of the following: An increase in symptoms, especially dyspnea or cough; An increase in opacities on chest CT scan, especially the development of honeycombing ; deterioration in lung function with > 10% decrease in FVC ( or > 200ml change) or > 15% decrease in DLCO (or at least > 3ml/min/mm Hg change).
- stable group: not included in improved group or deteriorated group

SUMMARY:
Diffuse Parenchymal Lung Disease(DPLD) is a chronic progressive fibrosis lung disease that with a highly variable clinical process.Krebs von den Lungen-6 (KL-6) is a high-molecular-weight glycoprotein, classified as human MUC1 mucin, that is produced mainly by regenerating type II pneumocytes.Serum levels of KL-6 have been shown to be elevated in patients with DPLD and could predict progress, but unaware of the differential threshold. The objective of this study was to perspectively and sequentially monitor serum KL-6 levels in patients with different DPLD,then analyze its clinical value and find the differential threshold.

DETAILED DESCRIPTION:
Subjects and Method: Recruiting different DPLD patients in our hospital between 2013 February and 2016 October, including polymyositis/dermatomyositis related interstitial lung disease (PM/DM-ILD), rheumatoid arthritis related interstitial lung disease (RA - ILD), interstitial pneumonia with autoimmune features(IPAF) and idiopathic pulmonary fibrosis(IPF), following up for enery 3 to 6 months. Once condition deteriorated, patient could return at any time if necessary according to our clinical physician judgment. Tumor markers，pulmonary function test(PFT); chest thin-section CT examination and CT scores; serum KL-6 levels were acquired in all patients at baseline and follow-ups. Serum KL-6 was measured on LUMIPULSE G System(FUJIREBIO, JAPAN) by chemiluminescence enzyme immunoassay. All follow-up patients will be respectively divided into improved,stable and deteriotated group according to the official ATS/ERS statement.

Inclusion criteria: (1)patient with PM/DM-ILD, RA-ILD, IPAF, IPF.The diagnosis of patient were according to the official ATS/ERS statement and the American College of Rheumatology/European League standard;(2)18 to 80 years old.

Exclusion criteria: (1)conbination with pulmonary tubenculersis,pulmonary infection,tumor;(2)no serum KL-6 or pulmonary function test or chest thin-section CT examintion ;(3)patient with severe hepatic and renal dysfunction,heart disease or receiving hemodialysis treatment;(4)pregnant or plan to be pregnant

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PM/DM-ILD,RA-ILD,IPAF,IPF

Exclusion Criteria:

* Combined with pulmonary infection,pulmonary tuberculosis,carsinoma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects with a dignosis of DPLD refer to the American Thracic Society(ATS)/European Respiratory Society(ERS) or American College of Rheumatology statement.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Serum KL-6 | 3 years
  serum samples were prospectively cellected from 180 patients at baseline and follow-ups. Serum KL-6 was measured on LUMIPULSE G System(FUJIREBIO, JAPAN) by chemiluminescence enzyme immunoassay.

SECONDARY OUTCOMES:
Forced vital capacity（FVC） | 3 years
  All patient were underwent spirometry examination on COSMED spirometer at baseline and follow-ups.Forced vital capacity（FVC）and the percentages of predicting value (FVC%pre) were recorded.
Diffusing capacity for carbon monoxide（DLCO） | 3 years
  All patient were underwent diffusion capacity examination by intra-breath method on COSMED spirometer at baseline and follow-ups.Diffusing capacity for carbon monoxide（DLCO）and the percentages of predicting value (DLCO%pre) were recorded.
CT score | 3 years
  All chest CT was obtained with 1 or 2 mm sequentially throughout the entire lung at baseline and follow-ups.CT scans were reviewed independtly by two thracic radiologists without knowledge of clinical,physiologic,or pathologic parameters,at a window level of -650 H and a window width of 1200 H. Obsevers were also kept unaware of patient diagnose.The whole lung were divided into six areas at the level of the aortic arch and inferior pulmonary vein.Each erea was scored on a scale of 0-10.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Guangzhou Medical university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No